CLINICAL TRIAL: NCT04138446
Title: Effects of Acute Hypobaric Hypoxia Exposure on Neurocognitive Performance of Pre-hospital Emergency Service Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Collaborators: Medical University Innsbruck (Other); University of Graz (Other); Università degli Studi di Trento (Other); Azienda Sanitaria dell'Alto Adige (Other); Istituto di Fisiologia Clinica CNR (Other)
Responsible Party: Principal Investigator, Giacomo Strapazzon, MD PhD, Principal Investigator, Institute of Mountain Emergency Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 3489044136
Record Dates: First submitted 2019-10-18; First posted 2019-10-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Hypobaric Hypoxia; Cognitive Deterioration; Emergency Medicine; Resuscitation; Stress Physiology

STUDY DESIGN:
Intervention Model Description: Interventional, non-pharmacological, randomized, controlled, single-blinded, cross-over
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 200-3000 (Experimental): Day 1: 200m (above sea level) asl Day 2: 3000m asl
  Interventions: Other: Altitude exposure in climate chamber
- 3000-200 (Experimental): Day 1: 3000m asl Day 2: 200m asl
  Interventions: Other: Altitude exposure in climate chamber
- 200-5000 (Experimental): Day 1: 200m asl Day 2: 5000m asl
  Interventions: Other: Altitude exposure in climate chamber
- 5000-200 (Experimental): Day 1: 5000m asl Day 2: 200m asl
  Interventions: Other: Altitude exposure in climate chamber
- 3000-5000 (Experimental): Day 1: 3000m asl Day 2: 5000m asl
  Interventions: Other: Altitude exposure in climate chamber
- 5000-3000 (Active Comparator): Day 1: 5000m asl Day 2: 3000m asl
  Interventions: Other: Altitude exposure in climate chamber

INTERVENTIONS:
Other: Altitude exposure in climate chamber — Altitude exposure in a climate chamber will consist of hypobaric hypoxia similar to the conditions found at 3000m asl and 5000m asl.

SUMMARY:
The study aims to evaluate the effects of acute hypobaric hypoxia on cognitive performance (H0: cognitive performance at 200 meters above sea level (asl) = cognitive performance at 3000 meters above sea level = cognitive performance at 5000 meters above sea level).

Before participating in the study, each participant will respond to a questionnaire related to high altitude exposure (prior 3 months), as well as inclusion/exclusion criteria evaluation.

On day 0, after the interview and signed informed consent, the participant will undergo a medical examination that will include a general objective examination. Participants will participate in a training on the emergency and safety procedures of the hypobaric hypoxia facility, as well as a refresh on cardiopulmonary resuscitation procedure.

During the following two days (day 1 and 2) the study protocol will be executed (one test per day). The study protocol envisages:

* a basal cognitive test battery
* blind ascent in the hypobaric chamber to simulated altitude
* cognitive test battery
* 5 minutes of recorded chest compressions on dummies
* cognitive test battery
* blind descent in the hypobaric chamber.

During the stay in the hypobaric hypoxic facility, each participant will be monitored in real time with the Equivital© medical monitoring device.

Before and after the stay in the hypobaric hypoxic facility, a saliva sample will be collected, and psychological tests administered.

ELIGIBILITY:
Inclusion criteria:

* Healthy volunteers
* Age 18-60 yr-old
* ASA class I
* Signed informed consent

Exclusion criteria:

* Age <18 or >60 yr-old
* ASA class > I
* Informed consent not signed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Digit-Symbol Substitution Task - DSST | Change from basal measurement (before altitude exposure) to altitude measurement (after altitude exposure - 5 minutes)
  Changes in working memory at altitude using a computer-based test (DSST)
Balloon Analog Risk Test - BART | Change from basal measurement (before altitude exposure) to altitude measurement (after altitude exposure - 5 minutes)
  Changes in risk-taking behavior at altitude using a computer-based test (BART)
Psychomotor Vigilance Test - PVT | Change from basal measurement (before altitude exposure) to altitude measurement (after altitude exposure - 5 minutes)
  Changes in reaction time using a computer-based test (PVT)

SECONDARY OUTCOMES:
Digit-Symbol Substitution Task - DSST | Change from rest measurement (altitude exposure before chest compressions) to post-exercise measurement (after 5 minutes of chest compressions at altitude)
  Changes in working memory after exercise at altitude using a computer-based test (DSST)
Balloon Analog Risk Test - BART | Change from rest measurement (altitude exposure before chest compressions) to post-exercise measurement (after 5 minutes of chest compressions at altitude)
  Changes in risk-taking behavior after exercise at altitude using a computer-based test (BART)
Psychomotor Vigilance Test - PVT | Change from rest measurement (altitude exposure before chest compressions) to post-exercise measurement (after 5 minutes of chest compressions at altitude)
  Changes in reaction time after exercise at altitude using a computer-based test battery (PVT)
Proportion of correct chest compressions regarding depth, pressure point and pressure release | Changes in 5 minute chest compressions
  Evaluation of the quality of chest compressions with a manikin and its electronic feedback device at different altitudes (200 meters vs. 3000 meters vs. 5000 meters)
Reactive oxygen species - ROS | Change from basal measurement (before altitude exposure) to post-altitude measurement (after altitude exposure - 1 hour)
  Changes in ROS in saliva samples (μmol/min)
Total antioxidant capacity - TAC | Change from basal measurement (before altitude exposure) to post-altitude measurement (after altitude exposure - 1 hour)
  Changes in TAC in saliva samples (mM)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Strapazzon, MD PhD, Principal Investigator — Eurac Research, Institute of Mountain Emergency Medicine
Locations (1):
- Eurac Research, Institute of Mountain Emergency Medicine, Bolzano, BZ, Italy

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months from study completion
Access Criteria: Access will be granted to primary collaborators who will be required to sign a Data Access agreement

REFERENCES:
- [Background] Taylor L, Watkins SL, Marshall H, Dascombe BJ, Foster J. The Impact of Different Environmental Conditions on Cognitive Function: A Focused Review. Front Physiol. 2016 Jan 6;6:372. doi: 10.3389/fphys.2015.00372. eCollection 2015. PMID 26779029
- [Background] Pietsch U, Strapazzon G, Ambuhl D, Lischke V, Rauch S, Knapp J. Challenges of helicopter mountain rescue missions by human external cargo: need for physicians onsite and comprehensive training. Scand J Trauma Resusc Emerg Med. 2019 Feb 13;27(1):17. doi: 10.1186/s13049-019-0598-2. PMID 30760298
- [Background] Li XY, Wu XY, Fu C, Shen XF, Yang CB, Wu YH. Effects of acute exposure to mild or moderate hypoxia on human psychomotor performance and visual-reaction time. Space Med Med Eng (Beijing). 2000 Aug;13(4):235-9. PMID 11892743
- [Background] Bouak F, Vartanian O, Hofer K, Cheung B. Acute Mild Hypoxic Hypoxia Effects on Cognitive and Simulated Aircraft Pilot Performance. Aerosp Med Hum Perform. 2018 Jun 1;89(6):526-535. doi: 10.3357/AMHP.5022.2018. PMID 29789086
- [Background] Basner M, Savitt A, Moore TM, Port AM, McGuire S, Ecker AJ, Nasrini J, Mollicone DJ, Mott CM, McCann T, Dinges DF, Gur RC. Development and Validation of the Cognition Test Battery for Spaceflight. Aerosp Med Hum Perform. 2015 Nov;86(11):942-52. doi: 10.3357/AMHP.4343.2015. PMID 26564759
- [Background] Wang JC, Tsai SH, Chen YL, Hsu CW, Lai KC, Liao WI, Li LY, Kao WF, Fan JS, Chen YH. The physiological effects and quality of chest compressions during CPR at sea level and high altitude. Am J Emerg Med. 2014 Oct;32(10):1183-8. doi: 10.1016/j.ajem.2014.07.007. Epub 2014 Jul 30. PMID 25154345
- [Derived] Vogele A, van Veelen MJ, Dal Cappello T, Falla M, Nicoletto G, Dejaco A, Palma M, Hufner K, Brugger H, Strapazzon G. Effect of Acute Exposure to Altitude on the Quality of Chest Compression-Only Cardiopulmonary Resuscitation in Helicopter Emergency Medical Services Personnel: A Randomized, Controlled, Single-Blind Crossover Trial. J Am Heart Assoc. 2021 Dec 7;10(23):e021090. doi: 10.1161/JAHA.121.021090. Epub 2021 Dec 2. PMID 34854317